CLINICAL TRIAL: NCT01145157
Title: A Comparison Between 'Signature™ Personalised Patient Care' to Conventional Total Knee Arthroplasty and Computer Assisted Navigation and a Cost Benefit Analysis for the Australian Market
Brief Title: A Comparison Between Signature Total Knee Arthroplasty (TKA) to Conventional TKA and Computer Assisted TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMET AU03 (INT.CR.LAU3)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Joint Disease
Keywords: knee; arthroplasty
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Signature Knee Guide (Experimental): Total Knee Arthroplasty using the Signature Knee Guide with the Vanguard Knee System
  Interventions: Device: Signature Knee Guide
- Conventional Instrumentation (Active Comparator): Total Knee Arthroplasty will be performed using Conventional Instrumentation with the Vanguard Knee System
  Interventions: Device: Conventional Instrumentation
- Computer Assisted Navigation (Active Comparator): Total Knee Arthroplasty will be performed using Computer Assisted Navigation with the Vanguard Knee System
  Interventions: Device: Computer Assisted Navigation

INTERVENTIONS:
Device: Signature Knee Guide — Total Knee Arthroplasty performed using Signature Knee Guide
  Arms: Signature Knee Guide
Device: Conventional Instrumentation — Total Knee Arthroplasty performed using Conventional Instrumentation
  Arms: Conventional Instrumentation
Device: Computer Assisted Navigation — Total Knee Arthroplasty performed using Computer Assisted Navigation
  Arms: Computer Assisted Navigation

SUMMARY:
This is a prospective, randomised clinical outcomes study comparing the Signature Personalised Patient Care, Conventional Total Knee Arthroplasty and Computer Assisted Navigation, using Vanguard Knee System. The aim of the study is to evaluate the safety and efficacy of TKA using Signature Personalised Patient Care compared to Conventional TKA and Computer Assisted Navigation.

DETAILED DESCRIPTION:
The objective of this study is to report and compare on the outcomes from patients undergoing total knee arthroplasty utilizing 'SignatureTM Personalised Patient Care', Conventional Total Knee Arthroplasty and Computer Assisted Navigation.

The 'SignatureTM Personalised Patient Care' is a system that uses a patient's Magnetic Resonance Imaging (MRI) and X-ray design to build surgical instruments customized for a patient's unique knee anatomy. Cutting positioning guides are produced to match the outer shape of the individual's distal femur and proximal tibia.

The cutting positioning guides are intended to be used as patient-specific surgical instrumentation to assist in the positioning of total knee replacement components intra-operatively and in guiding the marking of bone before cutting.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of legal age and skeletally mature
* Patient requires primary total knee arthroplasty due to non- inflammatory degenerative joint disease (e.g. osteoarthritis, traumatic arthritis, a vascular necrosis, dysplasia/DDH) or inflammatory joint disease (e.g., Rheumatoid arthritis).
* Patient has met an acceptable preoperative medical clearance and is free from or treated for cardiac, pulmonary, haematological, etc., conditions that would pose excessive operative risk
* The patient will be available for follow up throughout the duration of the study.

Exclusion Criteria:

* Patient is unable to have an MRI scan due to the following conditions:

  * Cardiac pacemaker
  * Surgical clips in head (aneurysm clips)
  * Some artificial heart valves
  * Electronic inner ear implants
  * Metal fragments in eyes
  * Electronic stimulators
  * Implanted pumps
* Patient has active infection or sepsis (treated or untreated)
* Patient has any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery.
* Patient is female of child-bearing age and not taking contraceptive precautions.
* Patient has inadequate bone stock to support the device (e.g. severe osteopenia, family history of severe osteoporosis or osteopenia).
* Patient has known moderate to severe renal insufficiency.
* Patient has a known or suspected metal sensitivity.
* Patient is immunosuppressed or receiving high doses of corticosteroids.
* Patient has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, or drug, alcohol abuse.
* Patient has BMI >40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Mechanical Axial Alignment | Six months post-operative
  The primary radiological outcome will be tibial rotation

SECONDARY OUTCOMES:
Functional outcomes - Knee Society Score | One year post-operative
  The Knee Score consists of points given for pain, range of motion, and stability in both the coronal and sagittal planes, with deductions for fixed deformity, and extensor lag. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.

CONTACTS AND LOCATIONS:
Overall Officials: Jegan Krishnan, Principal Investigator — Flinders Medical Centre
Locations (1):
- Repatriation General Hospital (RGH), Daw Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Patient Data

REFERENCES:
- [Derived] Cundy WJ, Theodoulou A, Ling CM, Krishnan J, Wilson CJ. Blood Loss in Total Knee Arthroplasty. J Knee Surg. 2017 Jun;30(5):452-459. doi: 10.1055/s-0036-1592147. Epub 2016 Sep 21. PMID 27652687